CLINICAL TRIAL: NCT01076114
Title: Comparison of Critical Flicker Fusion vs. Automated Visual Fields in the Detection of Early Glaucoma
Brief Title: Comparison of Critical Flicker Fusion Versus Automated Visual Fields in the Detection of Early Glaucoma
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Nassau University Medical Center (Other)
Responsible Party: Colin Scott, MD, Nassau University Medical Center
Other Study IDs: 09-320
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Patients with no evidence of glaucoma or as a suspect with normal intraocular pressure, normal cup to disc ratio with no other ocular pathology and a normal ophthalmic exam.
- Glaucoma Suspect: Patients with abnormal cup to disc ratio or increased intraocular pressure (>21mm/Hg) with an otherwise normal ophthalmic exam.

SUMMARY:
The purpose of this study is to evaluate if critical flicker fusion is a more reliable method for detection of early glaucoma compared to automated visual fields in comparison to subjects without evidence of glaucoma or optic nerve disease.

DETAILED DESCRIPTION:
Our hypothesis is that critical flicker fusion (CFF) is a more reliable method for detection of early glaucoma compared to automated visual fields in comparison to subjects without evidence of glaucoma or optic nerve disease. We aim to evaluate the structure of the optic nerve and compare it to results of visual fields and CFF. The CFF will also be correlated with intraocular pressure (IOP) measurements to observe if it may be more closely related than visual fields. This may become an additional tool to detect glaucoma in those with unreliable visual fields or who are unable to perform a visual field from physical or mental limitations.

ELIGIBILITY:
Inclusion:

* Glaucoma Suspects:
* Abnormal optic disc appearance with increased cup to disc ratio, or
* Increased intraocular pressure >21 in either eye
* Control Subjects:
* Normal appearing optic discs
* Normal intraocular pressure (<21)

Exclusion:

* Other ocular pathology
* History of seizures or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from routine clinic patients seen at the Eye Center at Nassau University Medical Center, in East Meadow, NY.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Difference of mean deviation of glaucoma suspects from controls between critical flicker fusion and automated visual fields. | 1 visit (1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Scott, MD, Principal Investigator — Nassau University Medical Center
Locations (1):
- Nassau University Medical Center, East Meadow, New York, United States

REFERENCES:
- [Background] Chen PC, Woung LC, Yang CF. Modulation transfer function and critical flicker frequency in high-myopia patients. J Formos Med Assoc. 2000 Jan;99(1):45-8. PMID 10743346
- [Background] Van Toi V, Grounauer PA, Burckhardt CW. Artificially increasing intraocular pressure causes flicker sensitivity losses. Invest Ophthalmol Vis Sci. 1990 Aug;31(8):1567-74. PMID 2387687
- [Background] Riddell LA. THE USE OF THE FLICKER PHENOMENON IN THE INVESTIGATION OF THE FIELD OF VISION. Br J Ophthalmol. 1936 Jul;20(7):385-410. doi: 10.1136/bjo.20.7.385. No abstract available. PMID 18169373
- [Background] Chang TT, Ciuffreda KJ, Kapoor N. Critical flicker frequency and related symptoms in mild traumatic brain injury. Brain Inj. 2007 Sep;21(10):1055-62. doi: 10.1080/02699050701591437. PMID 17891568
- [Background] Sharma P, Sharma BC, Tyagi P, Kumar M, Sarin SK. Neuropsychological impairment in severe acute viral hepatitis is due to minimal hepatic encephalopathy. Liver Int. 2009 Feb;29(2):260-4. doi: 10.1111/j.1478-3231.2008.01856.x. Epub 2008 Aug 14. PMID 18710429
- [Background] Patterson VH, Foster DH, Heron J, Mason RJ. Multiple sclerosis. Luminance threshold and measurements of temporal characteristics of vision. Arch Neurol. 1981 Nov;38(11):687-9. doi: 10.1001/archneur.1981.00510110047005. PMID 7305696
- [Background] Tyler CW. Specific deficits of flicker sensitivity in glaucoma and ocular hypertension. Invest Ophthalmol Vis Sci. 1981 Feb;20(2):204-12. PMID 7461923
- [Background] Yoshiyama KK, Johnson CA. Which method of flicker perimetry is most effective for detection of glaucomatous visual field loss? Invest Ophthalmol Vis Sci. 1997 Oct;38(11):2270-7. PMID 9344350
- [Background] Matsumoto C, Takada S, Okuyama S, Arimura E, Hashimoto S, Shimomura Y. Automated flicker perimetry in glaucoma using Octopus 311: a comparative study with the Humphrey Matrix. Acta Ophthalmol Scand. 2006 Apr;84(2):210-5. doi: 10.1111/j.1600-0420.2005.00588.x. PMID 16637839
- [Background] Tielsch JM, Sommer A, Katz J, Royall RM, Quigley HA, Javitt J. Racial variations in the prevalence of primary open-angle glaucoma. The Baltimore Eye Survey. JAMA. 1991 Jul 17;266(3):369-74. PMID 2056646
- [Background] Javitt JC, McBean AM, Nicholson GA, Babish JD, Warren JL, Krakauer H. Undertreatment of glaucoma among black Americans. N Engl J Med. 1991 Nov 14;325(20):1418-22. doi: 10.1056/NEJM199111143252005. PMID 1922253